CLINICAL TRIAL: NCT03478722
Title: Effect of Protein Ingestion on Postprandial Protein Handling in Hemodialysis Patients
Brief Title: Muscle Protein Synthesis in Dialysis Patients
Status: Completed | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Other Study IDs: 16203
Record Dates: First submitted 2018-03-19; First posted 2018-03-27 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-03

CONDITIONS: Muscle Loss
MeSH Terms: conditions — Muscular Atrophy | interventions — guar meal protein, Cyamopsis tetragonoloba

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma samples and skeletal muscle tissue biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Maintenance Hemodialysis Patients: Protein meal, stable isotope amino acid infusion
  Interventions: Other: Protein Meal; Other: Stable Isotope Amino Acid Infusion
- Control Subjects: Protein meal, stable isotope amino acid infusion
  Interventions: Other: Protein Meal; Other: Stable Isotope Amino Acid Infusion

INTERVENTIONS:
Other: Protein Meal — Ingestion of mixed meal containing 20 g of dietary protein
Other: Stable Isotope Amino Acid Infusion — Continuous infusion of L-[1-13C]leucine (0.13 μmol⋅kg⋅min) and L-[ring- 2H5]phenylalanine (0.05 μmol⋅kg⋅min)

SUMMARY:
The most severe form of chronic renal failure is end-stage-renal-disease with maintenance hemodialysis (MHD) as the most common treatment strategy. MHD patients experience a number of metabolic and phenotypic derangements including skeletal muscle wasting. Previously, it has been demonstrated that dialysis treatment leads to increased rates of forearm phenylalanine uptake (proxy for 'muscle' protein synthesis) with an even greater rates of phenylalanine release (proxy for 'muscle' protein breakdown). Hence, the dialysis procedure itself is catabolic and induces a catabolic carryover for several hours after dialysis. This suggests prolonged post-dialysis disturbances in whole body- and skeletal muscle protein metabolism in MHD patients. Moreover, dialysis treatment in itself results in ~20 % losses of circulating amino acids in the dialysate. Collectively, this creates the need for replacement of amino acids by protein supplementation during and/or after dialysis. The ingestion of protein-dense meals in between dialysis treatments likely represents an important dietary strategy to counterbalance dialysis-induced catabolism and to achieve the current recommended protein intakes (set at 1.2 g/kg bodyweight/d) to limit muscle protein loss in MHD patients. However, the effectiveness of protein-rich meal ingestion to augment postprandial whole body and muscle protein metabolic responses in MHD patients outside of the dialysis period remain largely undefined.

The purpose of this study is to compare basal and postprandial whole body leucine body kinetics, muscle anabolic sensing mechanisms, markers of muscle proteolysis, and myofibillar protein synthesis rates to mixed meal ingestion on a non-dialysis day in eight MHD patients, between 20-80 and to compare these outcomes to age- and BMI-matched controls. The investigators will use specifically produced intrinsically L-[5,5,5-2H3]leucine labeled eggs combined with primed constant amino acid tracer infusion methods and concomitant blood and muscle direct sampling to make direct assessments of in vivo protein digestion and absorption kinetics and subsequent postprandial muscle protein synthetic responses in MHD patents and controls. On the test day, subjects will remain sedentary for the determination of muscle protein synthesis in both the fasted state and after consumption of the meal.

DETAILED DESCRIPTION:
On the day of the infusion trial, participants will report to the laboratory at 0700 h after an overnight fast. MHD patients will be studied ~24 h after their dialysis treatment. A Teflon catheter will be inserted into an antecubital vein for baseline blood sample collection (t=-180 min) after which participants receive priming doses of NaH13CO2 (2.35 µmol·kg), L-[1-13C]leucine (7.6 µmol·kg FFM), and L-[ring-2H5]phenylalanine (2.0 µmol·kg FFM). Subsequently, a continuous intravenous infusion of L-[1-13C]leucine (0.10 µmol·kg FFM ·min) and L-[ring-2H5]phenylalanine (0.05 µmol·kg-1 FFM·min) will be initiated (t=-180 min) and maintained until the end of the trial. A second Teflon catheter will be inserted into a heated dorsal hand vein of the same arm for repeated arterialized blood sampling and will remain patent by a 0.9% saline drip. In the postabsorptive state, muscle biopsies will be collected at t=-120 and -0 min of the infusion. Subsequently, participants will consume a mixed meal containing 20 grams of dietary protein and the completion of the meal will mark the start of the postprandial phase (t=0 min). An additional muscle biopsy will be collected at 300 min to determine postprandial myofibrillar protein synthesis rates. Biopsies will be collected from the middle region of the vastus lateralis (15 cm above the patella) with a Bergström needle modified for suction under local anesthesia (2% Lidocaine). The postabsorptive muscle biopsies will be collected from the same incision with the needle pointed to distal and proximal directions, respectively. The postprandial biopsy will be collected through a separate incision 2-3 cm above the postabsorptive incision. All biopsy samples will be freed from any visible blood, adipose, and connective tissue immediately frozen in liquid nitrogen, and stored at -80˚C until subsequent analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-80 years (both healthy controls and MHD patients)
* Medical clearance from a Nephrologist at their respective dialysis clinic to participate (MHD patients)

Exclusion Criteria:

* Known allergies to egg consumption (both healthy controls and MHD patients)
* Phenylketonuria (both healthy controls and MHD patients)
* Vegans (both healthy controls and MHD patients)
* Diagnosed GI tract diseases (healthy controls)
* Recent (1 year) participation in amino acid tracer studies (both healthy controls and MHD patients)
* Predisposition to hypertrophic scarring or keloid formation (both healthy controls and MHD patients)
* Diabetes (healthy controls)
* Pregnancy (both healthy controls and MHD patients)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In total, the investigators would like to recruit 8 maintenance hemodialysis patients (both male and female) and 8 healthy controls matched for gender, age and BMI.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Fractional synthetic rate of myofibrillar proteins | 8 hours
  Measurement of muscle protein synthesis

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Burd, PhD, Principal Investigator — University of Illinois, Urbana-Champaign
Locations (1):
- Freer Hall, Urbana, Illinois, United States